CLINICAL TRIAL: NCT06229730
Title: Vestibular ASsessment In Children - Balance Function in Normal Children and Specific Risk Groups (VASIC)
Brief Title: Normative Data of Vestibular and Postural Function in Danish Children
Acronym: VASIC
Status: Recruiting | Type: Observational
Sponsor: Gødstrup Hospital (Other)
Responsible Party: Principal Investigator, Signe Fiil Bønløkke, Principal Investigator, Gødstrup Hospital
Other Study IDs: SFB-2-2023
Record Dates: First submitted 2024-01-08; First posted 2024-01-29 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Children, Only; Vestibular Function
Keywords: Vestibular dysfunction; Balance problem; Children; Dizziness; Vestibular assessment; video Head Impulse Test; Vestibular Evoked Myogenic Potential; Computerized Dynamic Posturography; Quality of life
MeSH Terms: conditions — Dizziness | interventions — Vestibular Evoked Myogenic Potentials

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy children without hearing or balance problems: Healthy children in the age of 6 months to 10 years, without any known hearing or balance problems and with normal gross motor development are recruited in local nurseries, kinder gardens, and schools.
  Interventions: Diagnostic Test: video Head Impulse Test; Diagnostic Test: Cervical Vestibular Evoked Myogenic Potential; Diagnostic Test: Ocular Vestibular Evoked Myogenic Potential; Diagnostic Test: Computerized Dynamic Posturography; Other: Dizziness Handicap Inventory for patient caregivers

INTERVENTIONS:
Diagnostic Test: video Head Impulse Test — For v-HIT, the Synapsys v-HIT Ulmer device is used.
  Other Names: vHIT
Diagnostic Test: Cervical Vestibular Evoked Myogenic Potential — For cVEMP, the Eclipse (Interacoustic, Middelfart, Denmark) is used. To bypass the frequent middle ear problems bone conduction stimuli (B-81, Interacoustic, Middelfart, Denmark) are administrated. The bone conductor is placed on the mastoid process and two trials at 70 dB nHL are conducted to check waveform reproducibility. 500 Hz short tone bursts (2-2-2 ms) are applied at 5 per second stimulus repetition rate.
  Other Names: cVEMP
Diagnostic Test: Ocular Vestibular Evoked Myogenic Potential — For oVEMP, the Eclipse (Interacoustic, Middelfart, Denmark) is used. To bypass the frequent middle ear problems bone conduction stimuli (B-81, Interacoustic, Middelfart, Denmark) are administrated. The bone conductor is placed on the mastoid process and two trials at 70 dB nHL are conducted to check waveform reproducibility. 500 Hz short tone bursts (2-2-2 ms) are applied at 5 per second stimulus repetition rate.
  Other Names: oVEMP
Diagnostic Test: Computerized Dynamic Posturography — To evaluate functional balance of the children and the relative contributions of the vision, proprioception, and vestibular system a CDP from Virtualis (Virtualis, Montpellier, France) is used.
  Other Names: CDP
Other: Dizziness Handicap Inventory for patient caregivers — DHI is a caregiver-reported 21-item questionnaire. It is designed to evaluate the perceived quality of life and handicap resulting from dizziness and unsteadiness for the pediatric population. For each question there are three possible answers: yes, sometimes or no. Each answer provides respectively 4, 2 and 0 points. The total DHI scores range from 0 to 84 with higher score being consistent with more limitation and more severe handicap. Scores under 16 are characterized as no limitation or handicap. A score from 16-26 present a mild perceived handicap and mild limitations. A DHI-score between 26-43 is classified as a moderate problem, and a score above 43 describes a severe perceived handicap and severe limitations.
  Other Names: DHI-PC

SUMMARY:
The goal of this age-based cohort study is to provide normative data of vestibular function in the general Danish pediatric population. Thus, the investigators will be able to compare patient data with norms, allowing for more precise diagnostics. The participants will be children in the age of 6 months to 10 years, without any known hearing or balance problems. The test protocol consists of questionnaires, hearing screening and vestibular and postural assessments.

DETAILED DESCRIPTION:
Balance problems in children are an overlooked issue in the Danish healthcare system. Dysfunction of the vestibular system, i.e. vestibular dysfunction (VD), can have significant consequences for children's development and quality of life.

Knowledge about the prevalence of vestibular impairment and normative data of vestibular function in the Danish pediatric population is missing.

The investigators aim for a child friendly and reliable vestibular test protocol in the study. According to the investigators studies as well as international reports, the investigators have chosen a vestibular test protocol with Video Head Impulse Test (v-HIT), cervical and ocular Vestibular Evoked Myogenic Potential (c and oVEMP) as the tests are feasible, valid, and child friendly. To evaluate overall balance ability, the children are tested on a Computerized Dynamic Posturography.

The aim of the study is to provide normative data of vestibular function in the general Danish pediatric population. Thus, the investigators will be able to compare patient data with norms, allowing for more precise diagnostics.

Methods: The study is an age-based cohort study. Participants are children in the age of 6 months to 10 years, without any known hearing or balance problems. The participants are recruited in local nurseries, kinder gardens, and schools. All participants will go through a test protocol consisting of questionnaires, hearing screening and vestibular and postural assessments.

The primary endpoints are age-based norms for v-HIT, c and oVEMP, and posturographic results. The secondary endpoints are number of subjects with successful results of the vestibular test protocol and mean total Dizziness Handicap Inventory for patient caregivers (DHI-PC) score. A number of variables are collected such as demographics, developmental milestones, family history with focus on hearing and balance.

ELIGIBILITY:
Inclusion Criteria:

* Children in the age of 6 months -10 years
* Normal hearing
* No history of dizziness or balance problems
* Written informed consent from the parents.

Exclusion Criteria:

* Premature birth
* Existing or previous inner ear disease(s) or previous inner ear surgery
* Cholesteatoma or previous middle ear surgery
* Known or previous vestibular disorder (Vestibular schwannoma, Mb Meniere, vestibular neuritis or other known)
* Delayed gross motor development evaluated through milestones.
* Visual impairment to such a degree that the child is not able to maintain fixation on a dot one meter away.
* Congenital nystagmus
* Compromised eye muscle mobility
* A diagnose of any neurological disease.
* A diagnose of any psychiatric disease.
* VEMP-electrode allergy
* History of symptomatic head or neck trauma
* Prescription of medicine which alters vestibular outputs (for instance sedative antihistamines)

Ages: 6 Months to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy children in the age of 6 months to 10 years, without any known hearing or balance problems (35 children in the age group from 6 months to 2 years, 30 children in the age group from 3 to 5 years, and 25 children from 6 to 10 years) are recruited in local nurseries, kinder gardens, and schools.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
video Head Impulse Test (vHIT) | Measured at baseline.
  Outcome measures: Age-based norms for mean VOR gain
video Head Impulse Test (vHIT) | Measured at baseline.
  Outcome measures: Age-based norms for VOR gain asymmetry in percent (%).
video Head Impulse Test (vHIT) | Measured at baseline.
  Outcome measures: Description of saccades (overt and covert saccades)
Cervical Vestibular Evoked Myogenic Potential (cVEMP): | Measured at baseline.
  Outcome measures: Age-based norms for latency P1 and latency N1 in milliseconds (ms)
Cervical Vestibular Evoked Myogenic Potential (cVEMP): | Measured at baseline.
  Outcome measures: Age-based norms for rectified interpeak amplitude P1-N1
Cervical Vestibular Evoked Myogenic Potential (cVEMP): | Measured at baseline.
  Outcome measures: Age-based norms for averaged EMG in µV
Cervical Vestibular Evoked Myogenic Potential (cVEMP): | Measured at baseline.
  Outcome measures: Age-based norms for left-right asymmetry ratio in percent (%)
Ocular Vestibular Evoked Myogenic Potential (oVEMP): | Measured at baseline.
  Outcome measures: Age-based norms for latency N1 and latency P1 in milliseconds
Ocular Vestibular Evoked Myogenic Potential (oVEMP): | Measured at baseline.
  Outcome measures: Age-based norms for interpeak amplitude N1-P1 in µV
Ocular Vestibular Evoked Myogenic Potential (oVEMP): | Measured at baseline.
  Outcome measures: Age-based norms for left-right asymmetry ratio in percent (%)
Computerized Dynamic Posturography (CDP) | Measured at baseline.
  Outcome measures: Aged-based norms for Sensory Organization Test (SOT):
  * Average equilibrium score (ES) for SOT1-6. Equilibrium scores is the average of three trials for each of the six conditions SOT1-6.
  * The SOT Composite score. It is a weighted average of the six conditions (SOT1-6) with greater weight given to the more difficult conditions.
  * The preference score. The preference score = (SOT3 + SOT6) / (SOT2 + SOT5)).
Computerized Dynamic Posturography (CDP) | Measured at baseline.
  Outcome measures: Aged-based norms for motor control test (MCT):
  • Mean latency of the medium and the big movement respectively in anterior and posterior direction measured in milliseconds.
Computerized Dynamic Posturography (CDP) | Measured at baseline.
  Outcome measures: Aged-based norms for adaptation test (ADT):
  • Mean sway energy score of toes-up and toes-down respectively. The sway energy score quantifies the force magnitude required to overcome the postural instability.

SECONDARY OUTCOMES:
Dizziness Handicap Inventory for patient caregivers (DHI-PC): | Measured at baseline.
  Outcome measures: Mean total DHI-PC score. DHI-PC is a caregiver-reported 21-item questionnaire. For each question there are three possible answers: yes, sometimes or no. Each answer provides respectively 4, 2 and 0 points. The total DHI scores range from 0 to 84 with higher score being consistent with more limitation and more severe handicap.
Success rate of the vestibular test protocol | Measured at baseline
  Number of subjects with successful results of each of the vestibular assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Therese Ovesen, Professor, Study Chair — University Clinic for Balance, Flavour and Sleep, Department of ENT, Gødstrup Hospital, DK
Locations (1):
- Gødstrup Regional Hospital, Herning, Denmark

IPD SHARING:
Plan to Share IPD: No